CLINICAL TRIAL: NCT06713525
Title: Copenhagen Pancreatic Cancer Study (COPAN)
Brief Title: Observational Copenhagen Pancreatic Cancer Study
Acronym: COPAN
Status: Not yet recruiting | Type: Observational
Sponsor: Inna Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Inna Chen, MD, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: PA2416
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with PC are referred to Comprehensive Pancreatic Cancer Center at Herlev Hospital

SUMMARY:
The primary objective of the Copenhagen Pancreatic Cancer (COPAN) study is to describe the real-world population of patients with pancreatic cancer (PC). Larger sample of longitudinal real-world data provides a unique opportunity for comprehensive exploration of the diagnostic and treatment journey for individuals diagnosed with PC and allows to investigate treatment outcomes and associated prognostic factors. Furthermore, the study aims to identify determinants of treatment management and treatment outcomes, including patient-reported outcomes.

DETAILED DESCRIPTION:
The study objective is to describe the real-world population of patients with pancreatic cancer by collecting longitudinal data that facilitates a more rigorous understanding of the PC. This research project will catalog different elements of a patient's diagnostic and treatment journey and identify unmet needs of patients with PC.

The study aims to:

1. To compile detailed demographic information of patients with PC.
2. To document and analyze the clinical and disease characteristics at the time of diagnosis and beyond.
3. To track various treatment modalities employed, including surgery, chemotherapy, and radiation therapy.
4. To assess short-term and long-term outcomes, including survival rates, complications, and quality of life.
5. To identify prognostic and predictive factors within the real-world cohort.

8. To investigate the impact of PC and treatment on patients' quality of life.

4 Study Design This study of patients with PC will employ both a prospective, observational design and retrospective design to capture real-world data relating to health status and/or the delivery of health care routinely collected from a variety of sources. Data will be collected longitudinally, allowing for a dynamic analysis of the disease trajectory.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed pancreatic cancer

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with pancreatic cancer referred to Department of Oncology, Herlev Hospital, Denmark within the study period will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

IPD SHARING:
Plan to Share IPD: No